CLINICAL TRIAL: NCT06161025
Title: A Phase 2/3, Multicenter, Randomized Study of Raludotatug Deruxtecan (R-DXd), a CDH6-directed Antibody-drug Conjugate, in Subjects With Platinum-resistant, High-grade Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study of Raludotatug Deruxtecan (R-DXd) in Subjects With Platinum-resistant, High-grade Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS6000-109; REJOICE-Ovarian01 (Other: Daiichi Sankyo); ENGOT-ov77 (Other: ENGOT); GOG-3096 (Other: GOG); jRCT2031230556 (Other: jRCT)
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Solid Cancer
Keywords: Primary pertioneal cancer; Ovarian cancer; Fallopian tube cancer; Raludotatug Deruxtecan (R-DXd); Cadherin 6 (CDH6)
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Topotecan; 1-dodecylpyridoxal; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: R-DXd 4.8mg/kg Q3W (Experimental): Participants will be randomized to receive intravenous R-DXd administered at a dose of 4.8 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: R-DXd
- Part A: R-DXd 5.6 mg/kg Q3W (Experimental): Participants will be randomized to receive intravenous R-DXd administered at a dose of 5.6 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: R-DXd
- Part A: R-DXd 6.4 mg/kg Q3W (Experimental): Participants will be randomized to receive intravenous R-DXd administered at a dose of 6.4 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: R-DXd
- Part B: R-DXd RP3D Q3W (Experimental): Participants will be randomized to receive intravenous R-DXd administered at the Recommended Phase 3 Dose (RP3D) every 3 weeks (Q3W).
  Interventions: Drug: R-DXd
- Part B: Investigator's Choice (Active Comparator): Participants will be randomized to receive intravenous treatment with investigator's choice of paclitaxel, pegylated liposomal doxorubicin (PLD), or topotecan.
  Interventions: Drug: Paclitaxel; Drug: Topotecan; Drug: PLD

INTERVENTIONS:
Drug: R-DXd — R-DXd will be administered as an intravenously (IV) infusion
  Other Names: DS-6000a
  Arms: Part A: R-DXd 4.8mg/kg Q3W; Part A: R-DXd 5.6 mg/kg Q3W; Part A: R-DXd 6.4 mg/kg Q3W; Part B: R-DXd RP3D Q3W
Drug: Paclitaxel — Paclitaxel will be administered as an IV infusion
  Arms: Part B: Investigator's Choice
Drug: Topotecan — Topotecan will be administered as an IV infusion
  Arms: Part B: Investigator's Choice
Drug: PLD — PLD will be administered as an IV infusion
  Other Names: Pegylated Liposomal Doxorubicin
  Arms: Part B: Investigator's Choice

SUMMARY:
This study will evaluate the safety and efficacy of R-DXd therapy in participants with ovarian, peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
This study will focus on R-DXd in participants with platinum-resistant, high-grade ovarian, primary peritoneal, or fallopian tube cancer. R-DXd is an antibody-drug conjugate that specifically binds to CDH6, which is overexpressed in tumor cells. The Phase 2 dose-optimization part of the study (Part A) intends to define the recommended dose based on safety and efficacy, while the Phase 3 (Part B) part of the study will compare R-DXd with Investigator's choice of chemotherapy and further evaluate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the informed consent form prior to the start of any study-specific qualification procedures.
* Age ≥18 years or the minimum legal adult age (whichever is greater) at the time the informed consent form is signed.
* Participants with histologically or cytologically documented high-grade serous ovarian cancer (OVC), high-grade endometrioid OVC, primary peritoneal cancer, or fallopian tube cancer.
* For Phase 2 (Part A) Participants must have at least 1 lesion, not previously irradiated, amenable to biopsy, and must consent to provide a pretreatment biopsy and on-treatment biopsy tissue sample (on-treatment biopsy sample not required for the Phase 3 part of the study). Fresh pretreatment biopsy may be waived for subjects who consent to provide an archival tumor tissue sample from a lesion not previously irradiated, performed within 6 months of consent and performed after treatment with their most recent cancer therapy regimen.
* For Phase 2 (Part A): Has received at least 1 but no more than 3 prior systemic lines of anticancer therapy. For Phase 3 (Part B): Has received at least 1 but no more than 4 prior systemic lines of anticancer therapy:

  * Neoadjuvant +/-adjuvant considered 1 line of therapy.
  * Maintenance therapy (eg, bevacizumab, poly-ADP ribose polymerase [PARP] inhibitors) will be considered part of the preceding line of therapy.
  * Therapy changed due to toxicity in the absence of progression will be considered part of the same line.
  * Hormonal therapy will be counted as a separate line of therapy, unless it was given as maintenance.
  * At least 1 line of therapy containing bevacizumab, unless the subject is not eligible for treatment with bevacizumab due to precautions/intolerance. Note: Subjects must have progressed radiologically on or after their most recent line of systemic therapy. Biochemical progression will not be considered progression for this study.
* Has platinum-resistant disease. If a subject had only 1 line of platinum therapy, must have received at least 4 cycles of platinum, must have had a best response of not PD, and then progressed between >90 and ≤180 days after the date of the last dose of platinum If a subject had 2 or 4 lines of platinum therapy, must have received at least 2 cycles of platinum and have progressed on or within 180 days after the date of the last dose of platinum.
* If mirvetuximab soravtansine (MIRV) is locally available: Has had prior treatment with MIRV for participants with documented high-folate receptor alpha expression, unless the participant is not eligible for treatment with mirvetuximab soravtansine due to precautions/intolerance, or if the treatment is not approved or available locally.
* Has at least 1 measurable lesion evaluated by computed tomography or magnetic resonance imaging according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) per investigator assessment.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Has adequate organ and bone marrow function as assessed by local laboratory (within 14 days before start of study drug administration).
* Is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures and study restrictions.
* For Phase 3 (Part B) only: Subjects must be eligible for one of the treatments included in the investigator's choice of chemotherapy arm.

Exclusion Criteria

* Has clear cell, mucinous, or sarcomatous histology, mixed tumors containing any histology, or low-grade/borderline OVC. (Note for Phase 3 [Part B]: seromucinous, low-grade serous carcinoma or ovarian sarcoma, carcinosarcoma and undifferentiated carcinoma are excluded.)
* Inadequate washout period before Cycle 1 Day 1, defined as follows:

  * Major surgery <28 days
  * Radiation therapy <28 days (if palliative stereotactic radiation therapy without abdominal radiation, ≤14 days)
  * Systemic anticancer therapy (including antibody-drug therapy, retinoid therapy, and hormonal therapy) <28 days or 5 half-lives, whichever is shorter, before starting study drug
  * Chloroquine/hydroxychloroquine <14 days
  * Exposure to another investigational drug within 28 days prior to start of study treatment or current participation in other therapeutic investigational procedures
* Clinically active brain metastases, spinal cord compression, or leptomeningeal carcinomatosis, defined as untreated or symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with untreated and asymptomatic brain metastases or subjects with treated brain metastases who are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy, at the investigator's discretion A minimum of 2 weeks must have elapsed between the end of radiotherapy and randomization and there should be no evidence of progression or need for steroid treatment or anticonvulsants for at least 2 weeks prior to randomization. Note: If there is a history or suspicion of central nervous system. Note: If there is a history or suspicion of central nervous system metastasis, a CT scan of the head or MRI of the brain must be performed at baseline.
* Any of the following within the past 6 months prior to randomization: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event.
* Uncontrolled or significant cardiovascular disease, including the following:

  * QT interval corrected with Fridericia's formula interval >470 ms.
  * Diagnosed or suspected long QT syndrome.
  * History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes.
  * The participant has bradycardia of less than 50 bpm, unless the subject has a pacemaker.
  * History of second- or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers and have no history of fainting or clinically relevant arrhythmia with pacemakers.
  * Myocardial infarction within 6 months prior to screening.
  * Uncontrolled angina pectoris within 6 months prior to screening.
  * New York Heart Association Class 3 or 4 congestive heart failure.
  * Left ventricular ejection fraction <50% or institutional lower limit of normal as measured by echocardiography or multigated acquisition (MUGA) scan.
  * Coronary/peripheral artery bypass graft within 6 months prior to screening
  * Uncontrolled hypertension (HgCTCAE Grade ≥3 hypertension as per NCI-CTCAE version 5.0).
  * Complete left or right bundle branch block.
* Has a history of (noninfectious) ILD/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion, etc) and any autoimmune, connective tissue, or inflammatory disorders with potential pulmonary involvement (eg, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc), or prior pneumonectomy.
* Chronic steroid treatment (>10 mg/day), with the exception of the following:

  * Inhaled steroids for asthma or COPD
  * Mineralocorticoids (eg, fludrocortisone) for subjects with orthostatic hypotension
  * Topical steroids for mild skin conditions
  * Low-dose supplemental corticosteroids for adrenocortical insufficiency
  * Premedication for treatment groups and/or premedication in case of any hypersensitivity
  * Intra-articular steroid injections
* History of malignancy other than epithelial OVC, primary peritoneal cancer, or fallopian tube cancer within 3 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (eg, 5-year OS rate >90%) and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, nonmelanoma skin carcinoma, ductal carcinoma in situ, or Stage 1 uterine cancer).
* Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE Version 5.0, Grade ≤1 or baseline. Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to Grade >2 for 3 months prior to randomization and managed with SOC treatment) that the investigator deems related to previous anticancer therapy, following discussion with the Sponsor, such as the following:

  * Chemotherapy-induced neuropathy
  * Fatigue
  * Endocrinopathies, which may include hypothyroidism, hyperthyroidism, Type 1 diabetes, hyperglycemia, and adrenal insufficiency
  * Skin pigmentation (vitiligo)
* For Phase 2 (Part A): Prior exposure to other CDH6-targeted agents or an ADC that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, trastuzumab deruxtecan or datopotamab deruxtecan). For Phase 3 (Part B): Prior exposure to other CDH6-targeted agents or an antibody-drug conjugate containing a topoisomerase I inhibitor.
* History of hypersensitivity to any excipients in the R-DXd or any known contraindication to treatment with, including hypersensitivity to, the study drug(s).
* Has an active or uncontrolled human immunodeficiency virus (HIV) infection.
* Has any evidence of severe or uncontrolled systemic diseases (including active bleeding diatheses or active infection, substance abuse) or other factors that, in the investigator's opinion, makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required.
* Has an active or uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Hepatitis B and Hepatitis C Screening tests are required.

Subjects are eligible if:

1. Hepatitis B virus surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
2. History of hepatitis C infection: eligible if the HCV viral load is below the level of detection in the absence of antiviral therapy during the previous 4 weeks.
3. Have normal transaminase values, or, if liver metastases are present, abnormal transaminases with a result of AST/ALT <3 × ULN, which are not attributable to HCV infection.

   * Female who is pregnant or breastfeeding or intends to become pregnant during the study.
   * Psychological, social, familial, or geographical factors that would prevent regular follow-up.
   * Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the subject; alter the absorption, distribution, metabolism, or excretion of the study drug; or confound the assessment of study results.
   * Has a history of receiving live-attenuated vaccine (messenger RNA [mRNA] and replication-deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first exposure to study intervention.
   * For Phase 3 (Part B) only: Has clinical symptoms or radiographic evidence of intestinal obstruction.
   * For Phase 3 (Part B) only: Has ascites or pleural effusions that require repeated drainage (less than 4 weeks between drainages).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Based on Blinded Independent Central Review (BICR) Assessment (Part A) | From date of randomization to data cut off, up to 18 months
  The ORR was defined as the percentage of participants with confirmed Complete Response (CR) or Partial Response (PR), by BICR assessment based on RECIST version 1.1.
Progression-free Survival (PFS) Based on BICR Assessment (Part B) | From date of randomization to data cut off, up to 26 months
  PFS is defined as the time from the date of randomization to the date of disease progression, defined as the first documented radiological progression or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Based on Investigator Assessment | From date of randomization to data cut off, up to 30 months
  The ORR was defined as the percentage of participants who achieved Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), by Investigator assessment based on RECIST version 1.1.
Overall Survival (OS) | From date of randomization to data cut off, up to 40 months
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Duration of Response (DOR) | From date of randomization to data cut off, up to 40 months
  DoR is defined as the time from the date of the first documentation of objective tumor response (CR or PR) that is subsequently confirmed to the first documentation of disease progression or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) Based on BICR and Investigator Assessment | From date of randomization to data cut off, up to 30 months
  PFS is defined as the time from the date of randomization to the date of disease progression, defined as the first documented radiological progression or death due to any cause.
Disease Control Rate (DCR) | From date of randomization to data cut off, up to 40 months
  DCR is defined as the proportion of participants who achieved a confirmed CR, PR, or stable disease maintained for ≥12 weeks, as assessed by BICR and investigator based on RECIST version 1.1
Time to Next Treatment (TTNT) | From date of randomization to data cut off, up to 40 months
  TTNT is defined as the time from randomization to the start date of the next line of therapy
Progression-free Survival 2 (PFS2) Based on Investigator Assessment | From date of randomization to data cut off, up to 40 months
  PFS2 is defined as the time from randomization to the first documented objective disease progression on next line therapy or death due to any cause, whichever comes first.
Percentage of Participants With Cancer Antigen 125 (CA-125) Response Rate | From baseline to data cut off, up to 40 months
  CA-125 response rate is defined as the percentage of participants with a reduction of 50% in CA-125 levels when compared to levels from a pretreatment sample, as assessed by blood sample based on Gynecological Cancer InterGroup criteria
Number of participants with Treatment-emergent Adverse Events (TEAEs) | From first dose to data cut off, up to 40 months
  TEAEs are defined as those AEs with a start or worsening date during the on-treatment period (from the first dose date to 40 days after the last dose date of study treatment).
Pharmacokinetic (PK) Analysis: Maximum Plasma Drug Concentration (Cmax) of R-DXd | From first dose to data cut off, up to 40 months
Pharmacokinetic (PK) Analysis: Time to Reach Maximum Plasma Drug Concentration (Tmax) of R-DXP | From first dose to data cut off, up to 40 months
Pharmacokinetic (PK) Analysis: Area Under the Concentration-Time Curve (AUC) of R-DXd | From first dose to data cut off, up to 40 months
Percentage of Participants With Treatment Emergent Antidrug Antibody (ADA) | From baseline to data cut off, up to 40 months
Pharmacokinetic (PK) Analysis: Terminal Half-Life (t1/2) of R-DXd | From first dose to data cut off, up to 40 months
Change from Baseline in Abdominal/gastrointestinal (GI) Symptoms (Part B) | From baseline to Week 12 and up to data cut off, up to 40 months
  Change from baseline in abdominal and gastrointestinal symptoms as measured by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) OV28 abdominal/GI subscale
Change from Baseline in Fatigue/Pain Symptoms (Part B) | From baseline to data cut off, up to 40 months
  Change from baseline as measured by the EORTC QLQ C30 Fatigue/Pain subscale score
Time to Deterioration in Fatigue/Pain Symptoms (Part B) | From baseline to data cut off, up to 40 months
  Time to deterioration in pain from baseline as measured by the EORTC QLQ C30 Fatigue/Pain subscale score
Time to Deterioration in GI Symptoms (Part B) | From baseline to data cut off, up to 40 months
  Time to deterioration in pain from baseline as measured by the EORTC QLQ OV28 abdominal/GI subscale total score
Time to Deterioration in Disease Impacts (Part B) | From baseline to data cut off, up to 40 months
  Time to deterioration in selected subscales of EORTC QLQ C30; physical functioning, global health status, overall quality of life.
Change from Baseline in Disease Impacts (Part B) | From baseline to data cut off, up to 40 months
  Change from Baseline in selected subscales of EORTC QLQ C30; physical functioning, global health status, overall quality of life.
Cadherin-6 (CDH6) protein expression in tumor tissue as determined by immunochemistry assay and correlation with ORR, DoR, PFS and OS | From baseline to data cut off, up to 40 months
  CDH6 protein expression in tumor tissue as determined by immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (120):
- United States (39):
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Yale University School of Medicine, New Haven, Connecticut
  - Sylvester Comprehensive Cancer Center at Lennar, Coral Gables, Florida
  - Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Florida Cancer Specialists, Lake Mary, Florida
  - Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Community MD Anderson Cancer Center- East, Indianapolis, Indiana
  - Community MD Anderson Cancer Center- South, Indianapolis, Indiana
  - Community Health Network - MD Anderson, Indianapolis, Indiana
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Washington University School of Medicine Obstetrics and Gynecology, St Louis, Missouri
  - Valley Health System, Paramus, New Jersey
  - Holy Name, Teaneck, New Jersey
  - NHPP Imbert, Bay Shore, New York
  - Northwell Health, LLC PRIME, Lake Success, New York
  - Perlmutter Cancer Center at NYU Langone Hospital- Long Island, Mineola, New York
  - NYU Langone Health, New York, New York
  - NHPP LHH, New York, New York
  - Duke Women's Cancer Care- Raleigh, Durham, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Ohio State University Wexner Medical Center, Hilliard, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Perelman School of Medicine at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sanford Cancer Center Gynecologic Oncology, Sioux Falls, South Dakota
  - Texas Oncology-Bedford, Bedford, Texas
  - Houston Area Locations- Woodlands, Conroe, Texas
  - Texas Oncology-Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology Paris, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas - MD Anderson, Houston, Texas
  - Houston Area Locations- Sugar Land, Houston, Texas
  - Houston Area Locations- West Houston, Houston, Texas
  - Houston Area Locations- League City, League City, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - GenesisCare St Andrews Hospital, Adelaide
  - GenesisCare North Shore (Oncology), St Leonards
- Canada (2):
  - McGill University Health Centre/Glen Site / Royal Victoria Hospital, Montreal
  - University Health Network - Princess Margaret Cancer Centre, Toronto
- China (13):
  - Beijing Cancer Hospital, Beijing
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Provincial Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Shandong Cancer Hospital, Jinan
  - Qilu Hospital of Shandong University, Jinan
  - Guangxi Medical University Cancer Hospital, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - National Cheng Kung University Hospital, Tainan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice v Motole, Prague
  - Fakultni nemocnice Bulovka, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (12):
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin - CLCC, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Groupe Hospitalier Diaconesses - Hôpital De La Croix Saint Simon, Paris
  - CARIO - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin
  - Institut Curie, Saint-Cloud
  - ICL Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (3):
  - Kliniken Essen-Mitte, Essen
  - Universitaetsklinikum Mannheim, Mannheim
  - Universitaetsklinikum Ulm, Ulm
- Italy (9):
  - IRCCS Centro di Riferimento Oncologico, Aviano
  - Azienda Ospedaliera Per Lemergenza Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Humanitas San Pio X, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale Mauriziano Umberto I, Torino
- Japan (12):
  - National Cancer Center Hospital, Chūōku
  - NHO Kyushu Cancer Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka-shi
  - National Cancer Center Hospital East, Kashiwa-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Jikei University Hospital, Minatoku
  - Shizuoka Cancer Center, Nagaizumi-cho
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Hokkaido University Hospital, Sapporo
  - Iwate Medical University Hospital, Shiwa-gun
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Mazowiecki Szpital Wojewodzki w Siedlcach Sp z o o, Siedlce
- Hospital Professor Doutor Fernando Fonseca, E.P.E., Amadora, Portugal
- South Korea (7):
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (9):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ciudad de Jaen, Jaén
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra (MAD), Pamplona
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clínico Universitario Valencia, Valencia
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan
- Royal United Hospital, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/